CLINICAL TRIAL: NCT00372671
Title: Evaluation of an Introductory Videotape Intervention to Improve Cardiac Rehabilitation Participation, the CR$P-2 Pilot Study.
Brief Title: Evaluation of an Introductory Videotape Intervention to Improve Cardiac Rehabilitation Participation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: R-02-144
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Myocardial Infarction; Unstable Angina; Coronary Angioplasty; Coronary Artery Bypass Surgery
Keywords: Cardiac Rehabilitation; Improving Cardiac Rehabilitation Participation
MeSH Terms: conditions — Myocardial Infarction; Angina, Unstable | interventions — Surveys and Questionnaires; Videotape Recording

INTERVENTIONS:
Behavioral: Survey
Behavioral: Survey and videotape

SUMMARY:
The purpose of this study is to determine whether a pre-discharge videotape introducing the concept and benefit of a Cardiac Rehabiliation & Secondary Prevention (CRSP) program will increase intent to participate in a CRSP program in post myocardial infarction, unstable angina, coronary artery bypass surgery, or coronary angioplasty patients.

DETAILED DESCRIPTION:
There is compelling evidence that a comprehensive CR program comprising the delivery of lifestyle modifying education will reduce mortality, morbidity and improve quality of life in patients following myocardial infarction, unstable angina, angioplasty or coronary artery bypass. However less than 20% of eligible patients participate in CRSP programs. This study will look at a method of potentially improving enrollment and adherence to a CRSP program. Patients will be randomized into two groups. One group will complete a survey and view a videotape introducing the concept of a CRSP program. The second group will be requested to complete a survey only, but will not be exposed to the videotape. It is expected that the patients who view the videotape will be more likely to express intent to participate in CRSP versus those patients who do not view the videotape.

ELIGIBILITY:
Inclusion Criteria:

* Admission to hospital for MI, UA, PTCA or CABS

Exclusion Criteria:

* Inability to provide written informed consent or complete the survey for any reason
* Previous CRSP participation
* Patients who are scheduled to undergo coronary artery bypass surgery within 3 months following the index hospital discharge
* Patients with an inability to exercise due to musculoskeletal problems or previous stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-06 (Actual); Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Expressed intent to participate in a CRSP program.

SECONDARY OUTCOMES:
Number of patients who continue to adhere to the 6-month CRSP program beyond the initial expressed intent to participate.
Impact of other patient variables and how they influence participation in a CRSP program.

CONTACTS AND LOCATIONS:
Overall Officials: Neville Suskin, MBChB, MSc, Principal Investigator — University of Western Ontario and London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada